CLINICAL TRIAL: NCT06413433
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Trial of Solriamfetol in Adults With Binge Eating Disorder (BED)
Brief Title: Elucidating TAAR-1, Dopamine, and Norepinephrine in Binge Eating Disorder Using Solriamfetol
Acronym: ENGAGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOL-BED-301
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Binge-Eating Disorder
Keywords: Binge eating disorder; BED; Solriamfetol; Sunosi; Axsome; Non-stimulant therapy; Dopamine norepinephrine reuptake inhibitor; Trace amine-associated receptor 1 (TAAR1) agonist
MeSH Terms: conditions — Binge-Eating Disorder | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Solriamfetol 150 mg (Experimental): Up to 12 weeks
  Interventions: Drug: Solriamfetol 150 mg
- Solriamfetol 300 mg (Experimental): Up to 12 weeks
  Interventions: Drug: Solriamfetol 300 mg
- Placebo (Placebo Comparator): Up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol 150 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 150 mg
Drug: Solriamfetol 300 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 300 mg
Drug: Placebo — Placebo tablets, taken once daily
  Arms: Placebo

SUMMARY:
ENGAGE (Elucidating TAAR-1, Dopamine, and Norepinephrine in Binge Eating Disorder Using Solriamfetol) is a Phase 3, randomized, double-blind, placebo-controlled, multicenter trial to assess the efficacy and safety of solriamfetol for the treatment of binge eating disorder (BED) in adults.

DETAILED DESCRIPTION:
Eligible subjects must have a diagnosis of BED according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria. Subjects will be randomized in a 1:1:1 ratio to receive solriamfetol (150 or 300 mg) or placebo, once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of BED according to DSM-5 criteria.
* Provides written informed consent to participate in the study before the conduct of any study procedures.
* Male or female, aged 18 to 55 inclusive.

Exclusion Criteria:

* Prior exposure to solriamfetol/Sunosi, through either a clinical study or prescription.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in number of binge eating episodes | 12 weeks

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Garden Grove, California
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Newport Beach, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, West Covina, California
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, Clermont, Florida
  - Clinical Research Site, Fort Myers, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lauderhill, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Marietta, Georgia
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Methuen, Massachusetts
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Princeton, New Jersey
  - Clinical Research Site, Mount Kisco, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Mason, Ohio
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, North Canton, Ohio
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Allentown, Pennsylvania
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Greenville, South Carolina
  - Clinical Research Site, North Charleston, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Draper, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com
- See also: ENGAGE Study Website — https://www.EngageBED.com